CLINICAL TRIAL: NCT05378659
Title: Neuroinflammation and Alzheimer's Pathology in Post-operative Cognitive Dysfunction: A Pilot Study
Brief Title: Neuroinflammation and Alzheimer's Pathology in POCD
Acronym: POCD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Other Study IDs: 4790
Record Dates: First submitted 2022-04-25; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Post-Operative Confusion; Neuroinflammatory Response; Alzheimer Disease
Keywords: POCD; Neuroinflammation
MeSH Terms: conditions — Alzheimer Disease; Neuroinflammatory Diseases | interventions — Mental Status and Dementia Tests; Stroop Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma and cerebrospinal fluid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With Post-Operative Cognitive Dysfunction: Subjects determined to have post-operative cognitive dysfunction based on the results of:
  1. 4AT Delirium Test
  2. Scoring on :
     1. Montreal Cognitive Assessment
     2. Oral Trails Test
     3. Stroop Test
     4. Symbol Digit Modalities Test
  All subjects will undergo:
  1. Blood sample collection
  2. Cerebral spinal fluid collection
  3. ERP testing
  4. NACC Cognitive Battery
  5. Grooved Pegboard testing
  Interventions: Behavioral: Montreal Cognitive Assessment; Behavioral: Stroop Test; Diagnostic Test: 4AT Delirium; Behavioral: Grooved Pegboard; Behavioral: NACC Cognitive Battery; Diagnostic Test: ERP Testing; Diagnostic Test: Blood Plasma and Serum sampling; Diagnostic Test: Cerebral Spinal Fluid Sample
- Without Post-Operative Cognitive Dysfunction: Subjects determined to not have post-operative cognitive dysfunction based on the results of:
  1. 4AT Delirium Test
  2. Scoring on :
     1. Montreal Cognitive Assessment
     2. Oral Trails Test
     3. Stroop Test
     4. Symbol Digit Modalities Test
  All subjects will undergo:
  1. Blood sample collection
  2. Cerebral spinal fluid collection
  3. ERP testing
  4. NACC Cognitive Battery
  5. Grooved Pegboard testing
  Interventions: Behavioral: Montreal Cognitive Assessment; Behavioral: Stroop Test; Diagnostic Test: 4AT Delirium; Behavioral: Grooved Pegboard; Behavioral: NACC Cognitive Battery; Diagnostic Test: ERP Testing; Diagnostic Test: Blood Plasma and Serum sampling; Diagnostic Test: Cerebral Spinal Fluid Sample

INTERVENTIONS:
Behavioral: Montreal Cognitive Assessment — Cognitive evaluation of short term memory, visuospatial abilities, executive functioning, attention, concentration, working memory, language, and orientation to time and place
  Other Names: MOCA
Behavioral: Stroop Test — Evaluates Processing Speed and Executive Control
Diagnostic Test: 4AT Delirium — Screening tool to test for delirium post surgery
Behavioral: Grooved Pegboard — Evaluation testing for dominant and non dominant sensory-motor speed
Behavioral: NACC Cognitive Battery — A series of tests that evaluate attention, concentration, immediate verbal memory, immediate visual memory, discrimination, processing/motor speed, and validity and effort.
Diagnostic Test: ERP Testing — An event-related potential ( ERP) is the measured brain response that is the direct result of a specific sensory, cognitive, or motor event. More formally, it is any stereotyped electrophysiological response to a stimulus. The study of the brain in this way provides a noninvasive means of evaluating brain functioning.
Diagnostic Test: Blood Plasma and Serum sampling — Up to six 4 ml samples of both serum and plasma will be obtained to assess for inflammatory markers.
Diagnostic Test: Cerebral Spinal Fluid Sample — At the time the spinal is placed for anesthetic purposes, 2ml of cerebral spinal fluid will be obtained to assess for inflammatory markers.

SUMMARY:
The purpose of this project is to investigate the role of both neural inflammation and pre-existing neurodegenerative pathology in the risk and pathogenesis of post-operative cognitive dysfunction (POCD). To achieve this goal, the investigators will combine blood and cerebrospinal fluid (CSF) sampling, standardized cognitive tests, and dynamic neurophysiological markers of cortical network dysfunction in the form of event-related potentials (ERPs), to assess the link between neurodegeneration and neuroinflammation in the pathogenesis of POCD.

DETAILED DESCRIPTION:
The purpose of this project is to investigate the role of both neural inflammation and pre-existing neurodegenerative pathology in the risk and pathogenesis of post-operative cognitive dysfunction (POCD) in 120 patients who will undergo a Total Knee Arthroscopy. The investigators will also explore neuropsychological, functional and biological measures as pre-operative risk indicators. To achieve this goal, the investigators will combine blood and cerebrospinal fluid (CSF) sampling, standardized cognitive tests, and dynamic neurophysiological markers of cortical network dysfunction in the form of event-related potentials (ERPs), to assess the link between neurodegeneration and neuroinflammation in the pathogenesis of POCD. To separate potential effects of general anesthesia from those of neuroinflammation, The investigators will recruit patients undergoing total knee replacement with the use of sedation and spinal anesthesia. To address the age risk factor, the investigators are targeting patients ages 60 and older. By using both validated and experimental biomarkers, this novel study design will isolate the effects of POCD due to systemic and neural inflammation and examine the links to pre-surgical cognitive impairment and underlying neurodegeneration as susceptibility factors.

Baseline (On the day of their final preoperative surgical visit prior to their TKA) the plan is to collect:

1. Cognitive assessments

   a. Montreal Cognitive Assessment b. Stroop Test c. Symbol Digit Modalities Test d. Oral Trail Making Test
2. Collect two 4-ml blood samples for biomarker evaluation

Visit 2 Pre-op (day of scheduled TKA surgery) the plan is to collect:

1. Repeat cognitive testing

   a. Montreal Cognitive Assessment b. Stroop Test c. Symbol Digit Modalities Test d. Oral Trail Making Test
2. Collect two 4-ml blood samples for biomarker evaluation
3. Collect 2cc of cerebral spinal fluid

Visit 2 Post-op:

1. 4 AT test for delirium
2. Collect two 4ml blood samples will be taken

Visit 3 (Forty-eight hours after discharge):

1. brief cognitive testing via telephone or video conferencing.

1. Blind Montreal Cognitive Assessment
2. Oral Trail Making Test

   Visit 4 (two weeks for their post-operative visit):

   1. Repeat cognitive testing

   1. Montreal Cognitive Assessment 2. Stroop Test 3. Symbol Digit Modalities Test 2. Oral Trail Making Test 3. Collect two 4ml blood samples for biomarker testing.

   For patients who had pre-operative cognitive impairment, their participation in the study will end here

   For 20 participants with no indication of pre-surgical cognitive impairment (10 with no post-operative impairment and 10 with presumed POCD)

   Visit 5 (~ 6 weeks post-op) the plan is to collect:
   1. Complete initial neurophysiological recording of event-related potentials (ERPs). This ERP session is performed to establish baseline cortical network function. Neurophysiological studies will be conducted using a 128-electrode EEG system.
   2. Collect two 4-ml blood samples

   Visit 6 End of Study (At 6 months):
   1. Collect a final assessment of cognition
   2. ERP assessment

ELIGIBILITY:
Inclusion Criteria:

* Males and females 60 years or older in age
* Subjects scheduled to undergo TKA
* Fluent and literate in English
* Able to give consent for themselves based upon the MacArthur Competence Assessment Tool for Clinical Research
* Able to have a subarachnoid block with only intravenous sedation

Exclusion Criteria:

* Less than 60 years of age
* Cognitively impaired to the point where they are unable to give consent for themselves
* Blindness or partial blindness
* Pre-existing neurodegenerative conditions
* Contraindication for subarachnoid block and/or requiring general anesthesia

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: No one ethnic group is either targeted or excluded in the proposed study. The investigators aim to target a sample of individuals ages 60 and older who will all undergo total knee arthroplasty. This selection of participants is based upon the aims of the current study.
  Due to the nature of the study, the investigators will include individuals with who are considered elderly. This population is necessary due to the increased prevalence of POCD within this group.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Blood Interleukin-1 beta (IL-1β) | Baseline
  A proinflammatory cytokine that activates astrocytes and micro ganglia
Blood Interleukin-1 beta (IL-1β) | Pre-op (pre-operation) -Visit 2- Day of surgery
  A proinflammatory cytokine that activates astrocytes and micro ganglia
Blood Interleukin-1 beta (IL-1β) | Post-op Visit 2- In recovery room up to 12 hours post surgery
  A proinflammatory cytokine that activates astrocytes and micro ganglia
Blood Interleukin-1 beta (IL-1β) | 2 Week Post-op -Visit 4
  A proinflammatory cytokine that activates astrocytes and micro ganglia
Blood Interleukin-1 beta (IL-1β) | 6 Week Post-op -Visit 5
  A proinflammatory cytokine that activates astrocytes and micro ganglia
Blood Tumor necrosis factor alpha (TNF- α) | Baseline
  A proinflammatory cytokine associated with neuroinflammation associated with neurodegenerative diseases
Blood Tumor necrosis factor alpha (TNF- α) | Pre-op- Visit 2- Day of surgery
  A proinflammatory cytokine associated with neuroinflammation associated with neurodegenerative diseases
Blood Tumor necrosis factor alpha (TNF- α) | Post-op Visit 2- In recovery room up to 12 hours post surgery
  A proinflammatory cytokine associated with neuroinflammation associated with neurodegenerative diseases
Blood Tumor necrosis factor alpha (TNF- α) | 2-week Post-op Visit 4
  A proinflammatory cytokine associated with neuroinflammation associated with neurodegenerative diseases
Blood Tumor necrosis factor alpha (TNF- α) | 6-week Post-op Visit 5
  A proinflammatory cytokine associated with neuroinflammation associated with neurodegenerative diseases
Blood Macrophage inflammatory protein-1 alpha (MIP-1alpha) | Baseline
  A chemotactic cytokine which plays a role in the inflammatory process of Alzheimer's Disease
Blood Macrophage inflammatory protein-1 alpha (MIP-1alpha) | Pre-op Visit 2- Day of surgery
  A chemotactic cytokine which plays a role in the inflammatory process of Alzheimer's Disease
Blood Macrophage inflammatory protein-1 alpha (MIP-1alpha) | Post-op Visit 2- In recovery room up to 12 hours post surgery
  A chemotactic cytokine which plays a role in the inflammatory process of Alzheimer's Disease
Blood Macrophage inflammatory protein-1 alpha (MIP-1alpha) | 2-week Post-op Visit 4
  A chemotactic cytokine which plays a role in the inflammatory process of Alzheimer's Disease
Blood Macrophage inflammatory protein-1 alpha (MIP-1alpha) | 6- week Post-op Visit 5
  A chemotactic cytokine which plays a role in the inflammatory process of Alzheimer's Disease
Blood Monocyte chemoattractant protein-1 (MCP-1/CCL2) | Baseline
  A chemotactic cytokine which plays a role in the inflammatory process through the regulation of monocytes/macrophages
Blood Monocyte chemoattractant protein-1 (MCP-1/CCL2) | Pre-op Visit 2- Day of surgery
  A chemotactic cytokine which plays a role in the inflammatory process through the regulation of monocytes/macrophages
Blood Monocyte chemoattractant protein-1 (MCP-1/CCL2) | Post-op Visit 2- In recovery room up to 12 hours post surgery
  A chemotactic cytokine which plays a role in the inflammatory process through the regulation of monocytes/macrophages
Blood Monocyte chemoattractant protein-1 (MCP-1/CCL2) | 2 week Post-op Visit 4
  A chemotactic cytokine which plays a role in the inflammatory process through the regulation of monocytes/macrophages
Blood Monocyte chemoattractant protein-1 (MCP-1/CCL2) | 6 week- Post-op Visit 5
  A chemotactic cytokine which plays a role in the inflammatory process through the regulation of monocytes/macrophages
Cerebral Spinal Fluid Phosphorylated Tau Protein | Pre-op Visit 2-Day of surgery
  A helical protein known to be a biomarker in the cerebral spinal fluid in brains with Alzheimer's Disease
ERP response amplitude | 6 Week post-op visit 5
  Measurement of event related potentials in the brain
ERP response latency | 6 Week post-op visit 5
  Measurement of event related potentials in the brain
ERP response amplitude | 6 Month post-op visit 6
  Measurement of event related potentials in the brain
ERP response latency | 6 Month post-op visit 6
  Measurement of event related potentials in the brain
Stroop Test | Baseline
  A neurocognitive test used to assess cognitive interference. T-Scores are computed with scores above 40 being "normal."
Stroop Test | Pre-op Visit 2- Day of surgery
  A neurocognitive test used to assess cognitive interference. T-Scores are computed with scores above 40 being "normal."
Stroop Test | 2 Week post-op Visit 4
  A neurocognitive test used to assess cognitive interference. T-Scores are computed with scores above 40 being "normal."
Montreal Cognitive Assessment | Baseline
  A neurocognitive test used to assess cognitive function across multiple domains. Scoring is on a scale from 0-30 with a score >26 being normal.
Montreal Cognitive Assessment | Pre-op Visit 2- Day of surgery
  A neurocognitive test used to assess cognitive function across multiple domains. Scoring is on a scale from 0-30 with a score >26 being normal.
Blind Montreal Cognitive Assessment | 48 Hours post-op- Visit 3
  A neurocognitive test used to assess cognitive function across multiple domains. Scoring is on a scale from 0-22 with a score >18 being normal.
Montreal Cognitive Assessment | 2 Week post-op- Visit 4
  A neurocognitive test used to assess cognitive function across multiple domains. Scoring is on a scale from 0-30 with a score >26 being normal.
Oral Trail Making Test | Baseline
  A neurocognitive test used to assess cognitive executive function with times for trail A > 78 seconds and trail B >273 seconds being deficient.
Oral Trail Making Test | Pre-op Visit 2- Day of surgery
  A neurocognitive test used to assess cognitive executive function with times for trail A > 78 seconds and trail B >273 seconds being deficient.
Oral Trail Making Test | 48 Hours post-op Visit 3
  A neurocognitive test used to assess cognitive executive function with times for trail A > 78 seconds and trail B >273 seconds being deficient.
Oral Trail Making Test | 2- Week post-op Visit 4
  A neurocognitive test used to assess cognitive executive function with times for trail A > 78 seconds and trail B >273 seconds being deficient.
Symbol Digit Test | Baseline
  A neurocognitive test used to assess for cerebral dysfunction scored through statistical methods with a higher score meaning higher cognitive vitality.
Symbol Digit Test | Pre-op Visit 2- Day of surgery
  A neurocognitive test used to assess for cerebral dysfunction scored through statistical methods with a higher score meaning higher cognitive vitality.
Symbol Digit Test | 2- Week post-op Visit 4
  A neurocognitive test used to assess for cerebral dysfunction scored through statistical methods with a higher score meaning higher cognitive vitality.
4 AT Delirium Screening | Post-op Visit 2- In recovery room up to 12 hours post surgery
  Bedside screening to detect delirium with a score of 4 or more indicating delirium +/- cognitive impairment, and a score of 1-3 indicating possible cognitive impairment.
Grooved Pegboard Test | 6 month post-op Visit 6
  A neurocognitive test consisting of varying key shapes and matching holes used to test visual motor coordination with a higher score indicating less or no impairment based on the individual's age and sex.
National Alzheimer's Coordinating Center Cognitive Battery | 6 month post-op Visit 6
  Cognitive assessment to test for deficits across multiple domains with a score of 95/995 =physical problem; 96/996 = cognitive/behavioral problem

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Craft, MD, Principal Investigator — University of Tennessee Graduate School of Medicine
Locations (1):
- Robert M Craft, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators who proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- [Background] Daiello LA, Racine AM, Yun Gou R, Marcantonio ER, Xie Z, Kunze LJ, Vlassakov KV, Inouye SK, Jones RN, Alsop D, Travison T, Arnold S, Cooper Z, Dickerson B, Fong T, Metzger E, Pascual-Leone A, Schmitt EM, Shafi M, Cavallari M, Dai W, Dillon ST, McElhaney J, Guttmann C, Hshieh T, Kuchel G, Libermann T, Ngo L, Press D, Saczynski J, Vasunilashorn S, O'Connor M, Kimchi E, Strauss J, Wong B, Belkin M, Ayres D, Callery M, Pomposelli F, Wright J, Schermerhorn M, Abrantes T, Albuquerque A, Bertrand S, Brown A, Callahan A, D'Aquila M, Dowal S, Fox M, Gallagher J, Anna Gersten R, Hodara A, Helfand B, Inloes J, Kettell J, Kuczmarska A, Nee J, Nemeth E, Ochsner L, Palihnich K, Parisi K, Puelle M, Rastegar S, Vella M, Xu G, Bryan M, Guess J, Enghorn D, Gross A, Gou Y, Habtemariam D, Isaza I, Kosar C, Rockett C, Tommet D, Gruen T, Ross M, Tasker K, Gee J, Kolanowski A, Pisani M, de Rooij S, Rogers S, Studenski S, Stern Y, Whittemore A, Gottlieb G, Orav J, Sperling R; SAGES Study Group*. Postoperative Delirium and Postoperative Cognitive Dysfunction: Overlap and Divergence. Anesthesiology. 2019 Sep;131(3):477-491. doi: 10.1097/ALN.0000000000002729. PMID 31166241
- [Background] O' Brien H, Mohan H, Hare CO, Reynolds JV, Kenny RA. Mind Over Matter? The Hidden Epidemic of Cognitive Dysfunction in the Older Surgical Patient. Ann Surg. 2017 Apr;265(4):677-691. doi: 10.1097/SLA.0000000000001900. PMID 27537541
- [Background] Chen MH, Liao Y, Rong PF, Hu R, Lin GX, Ouyang W. Hippocampal volume reduction in elderly patients at risk for postoperative cognitive dysfunction. J Anesth. 2013 Aug;27(4):487-92. doi: 10.1007/s00540-012-1548-6. Epub 2013 Jan 31. PMID 23371369
- [Background] Pappa M, Theodosiadis N, Tsounis A, Sarafis P. Pathogenesis and treatment of post-operative cognitive dysfunction. Electron Physician. 2017 Feb 25;9(2):3768-3775. doi: 10.19082/3768. eCollection 2017 Feb. PMID 28465805
- [Background] Xiao QX, Liu Q, Deng R, Gao ZW, Zhang Y. Postoperative cognitive dysfunction in elderly patients undergoing hip arthroplasty. Psychogeriatrics. 2020 Jul;20(4):501-509. doi: 10.1111/psyg.12516. Epub 2020 Jan 24. PMID 31976614
- [Background] Feinkohl I, Winterer G, Spies CD, Pischon T. Cognitive Reserve and the Risk of Postoperative Cognitive Dysfunction. Dtsch Arztebl Int. 2017 Feb 17;114(7):110-117. doi: 10.3238/arztebl.2017.0110. PMID 28302254
- [Background] Evered L, Scott DA, Silbert B, Maruff P. Postoperative cognitive dysfunction is independent of type of surgery and anesthetic. Anesth Analg. 2011 May;112(5):1179-85. doi: 10.1213/ANE.0b013e318215217e. Epub 2011 Apr 7. PMID 21474666
- [Background] Mason SE, Noel-Storr A, Ritchie CW. The impact of general and regional anesthesia on the incidence of post-operative cognitive dysfunction and post-operative delirium: a systematic review with meta-analysis. J Alzheimers Dis. 2010;22 Suppl 3:67-79. doi: 10.3233/JAD-2010-101086. PMID 20858956
- [Background] Edipoglu IS, Celik F. The Associations Between Cognitive Dysfunction, Stress Biomarkers, and Administered Anesthesia Type in Total Knee Arthroplasties: Prospective, Randomized Trial. Pain Physician. 2019 Sep;22(5):495-507. PMID 31561651
- [Background] Bekker A, Lee C, de Santi S, Pirraglia E, Zaslavsky A, Farber S, Haile M, de Leon MJ. Does mild cognitive impairment increase the risk of developing postoperative cognitive dysfunction? Am J Surg. 2010 Jun;199(6):782-8. doi: 10.1016/j.amjsurg.2009.07.042. PMID 20609722
- [Background] Silbert B, Evered L, Scott DA, McMahon S, Choong P, Ames D, Maruff P, Jamrozik K. Preexisting cognitive impairment is associated with postoperative cognitive dysfunction after hip joint replacement surgery. Anesthesiology. 2015 Jun;122(6):1224-34. doi: 10.1097/ALN.0000000000000671. PMID 25859906
- [Background] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Background] Luo A, Yan J, Tang X, Zhao Y, Zhou B, Li S. Postoperative cognitive dysfunction in the aged: the collision of neuroinflammaging with perioperative neuroinflammation. Inflammopharmacology. 2019 Feb;27(1):27-37. doi: 10.1007/s10787-018-00559-0. Epub 2019 Jan 3. PMID 30607668
- [Background] Simen AA, Bordner KA, Martin MP, Moy LA, Barry LC. Cognitive dysfunction with aging and the role of inflammation. Ther Adv Chronic Dis. 2011 May;2(3):175-95. doi: 10.1177/2040622311399145. PMID 23251749
- [Background] Ortega-Gomez A, Perretti M, Soehnlein O. Resolution of inflammation: an integrated view. EMBO Mol Med. 2013 May;5(5):661-74. doi: 10.1002/emmm.201202382. Epub 2013 Apr 17. PMID 23592557
- [Background] Ferretti MT, Cuello AC. Does a pro-inflammatory process precede Alzheimer's disease and mild cognitive impairment? Curr Alzheimer Res. 2011 Mar;8(2):164-74. doi: 10.2174/156720511795255982. PMID 21345170
- [Background] Meraz-Rios MA, Toral-Rios D, Franco-Bocanegra D, Villeda-Hernandez J, Campos-Pena V. Inflammatory process in Alzheimer's Disease. Front Integr Neurosci. 2013 Aug 13;7:59. doi: 10.3389/fnint.2013.00059. eCollection 2013. PMID 23964211
- [Background] Hu Z, Ou Y, Duan K, Jiang X. Inflammation: a bridge between postoperative cognitive dysfunction and Alzheimer's disease. Med Hypotheses. 2010 Apr;74(4):722-4. doi: 10.1016/j.mehy.2009.10.040. Epub 2009 Nov 26. PMID 19944539
- [Background] Andreasen N, Hesse C, Davidsson P, Minthon L, Wallin A, Winblad B, Vanderstichele H, Vanmechelen E, Blennow K. Cerebrospinal fluid beta-amyloid(1-42) in Alzheimer disease: differences between early- and late-onset Alzheimer disease and stability during the course of disease. Arch Neurol. 1999 Jun;56(6):673-80. doi: 10.1001/archneur.56.6.673. PMID 10369305
- [Background] Evered L, Silbert B, Scott DA, Ames D, Maruff P, Blennow K. Cerebrospinal Fluid Biomarker for Alzheimer Disease Predicts Postoperative Cognitive Dysfunction. Anesthesiology. 2016 Feb;124(2):353-61. doi: 10.1097/ALN.0000000000000953. PMID 26580833
- [Background] Wu Z, Zhang M, Zhang Z, Dong W, Wang Q, Ren J. Ratio of beta-amyloid protein (Abeta) and Tau predicts the postoperative cognitive dysfunction on patients undergoing total hip/knee replacement surgery. Exp Ther Med. 2018 Jan;15(1):878-884. doi: 10.3892/etm.2017.5480. Epub 2017 Nov 10. PMID 29399093
- [Background] Xie Z, McAuliffe S, Swain CA, Ward SA, Crosby CA, Zheng H, Sherman J, Dong Y, Zhang Y, Sunder N, Burke D, Washicosky KJ, Tanzi RE, Marcantonio ER. Cerebrospinal fluid abeta to tau ratio and postoperative cognitive change. Ann Surg. 2013 Aug;258(2):364-9. doi: 10.1097/SLA.0b013e318298b077. PMID 23732272
- [Background] Shi HJ, Xue XH, Wang YL, Zhang WS, Wang ZS, Yu AL. Effects of different anesthesia methods on cognitive dysfunction after hip replacement operation in elder patients. Int J Clin Exp Med. 2015 Mar 15;8(3):3883-8. eCollection 2015. PMID 26064288
- [Background] Gaetani L, Blennow K, Calabresi P, Di Filippo M, Parnetti L, Zetterberg H. Neurofilament light chain as a biomarker in neurological disorders. J Neurol Neurosurg Psychiatry. 2019 Aug;90(8):870-881. doi: 10.1136/jnnp-2018-320106. Epub 2019 Apr 9. PMID 30967444
- [Background] Niikado M, Chrem-Mendez P, Itzcovich T, Barbieri-Kennedy M, Calandri I, Martinetto H, Serra M, Calvar J, Campos J, Russo MJ, Pertierra L, Allegri R, Sevlever G, Surace EI. Evaluation of Cerebrospinal Fluid Neurofilament Light Chain as a Routine Biomarker in a Memory Clinic. J Gerontol A Biol Sci Med Sci. 2019 Mar 14;74(4):442-445. doi: 10.1093/gerona/gly179. PMID 30107413
- [Background] Frisoni GB, Fox NC, Jack CR Jr, Scheltens P, Thompson PM. The clinical use of structural MRI in Alzheimer disease. Nat Rev Neurol. 2010 Feb;6(2):67-77. doi: 10.1038/nrneurol.2009.215. PMID 20139996
- [Background] Galvao-Carmona A, Gonzalez-Rosa JJ, Hidalgo-Munoz AR, Paramo D, Benitez ML, Izquierdo G, Vazquez-Marrufo M. Disentangling the attention network test: behavioral, event related potentials, and neural source analyses. Front Hum Neurosci. 2014 Oct 13;8:813. doi: 10.3389/fnhum.2014.00813. eCollection 2014. PMID 25352800
- [Background] McMackin R, Bede P, Pender N, Hardiman O, Nasseroleslami B. Neurophysiological markers of network dysfunction in neurodegenerative diseases. Neuroimage Clin. 2019;22:101706. doi: 10.1016/j.nicl.2019.101706. Epub 2019 Feb 2. PMID 30738372